CLINICAL TRIAL: NCT00298298
Title: L-Vax: A Feasibility Study Using a DNP-Modified Autologous Tumor Cell Vaccine as Therapy in Patients With Resectable Non-Small Cell Lung Cancer
Brief Title: DNP-Modified Autologous Tumor Cell Vaccine for Resectable Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Suspended until capitalization is completed
Sponsor: AVAX Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A/100/0601
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Non-Small Cell Lung Cancer - Completely Resectable
Keywords: lung cancer; non-small cell lung cancere; vaccine; immunotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 5 million autologous, DNP-modified NSCLC cells
  Interventions: Biological: L-Vax: Autologous, DNP-Modified NSCLC Vaccine
- 2 (Experimental): 2.5 million autologous, DNP-modified NSCLC cells
  Interventions: Biological: L-Vax: Autologous, DNP-Modified NSCLC Vaccine
- 3 (Experimental): 0.5 million autologous, DNP-modified NSCLC cells
  Interventions: Biological: L-Vax: Autologous, DNP-Modified NSCLC Vaccine

INTERVENTIONS:
Biological: L-Vax: Autologous, DNP-Modified NSCLC Vaccine — autologous, DNP-modified NSCLC cells in suspension dosage - depends on arm route - intradermal frequency - weekly x7, booster at 6 months

SUMMARY:
To determine if a vaccine made from patient's own tumor tissue can stimulate an immune response against the patient's tumor cells. To determine the safety of the vaccine

DETAILED DESCRIPTION:
Study Objectives: To study the toxicity, safety and delayed-type hypersensitivity (DTH) responses of DNP-modified autologous tumor cell vaccine (L-Vax) in patients with resectable NSCLC:

* To determine the tolerability and toxicity of L-Vax
* To determine whether L-Vax induces a DTH response to autologous, DNP-modified NSCLC cells of similar magnitude to responses observed with melanoma
* Determine whether L-Vax induces a DTH response to autologous unmodified NSCLC cells
* To determine whether the DTH responses to autologous, unmodified NSCLC cells that have been fixed with ethanol correlate with DTH responses to autologous, unmodified NSCLC cells that are not fixed

Study Population: Patients with resectable NSCLC whose therapeutic tumor surgery provides a mass, which yields adequate tumor, cells for vaccine preparation and DTH testing

Study Design: A Phase I/IIa double-blind, three-dose, single center study

Investigational Product: L-Vax: DNP-modified autologous NSCLC cell vaccine

Dosage Form: Cell suspension

Route of Administration: Intradermal

Dosage and Treatment Schedule: Prior to vaccine administration, patients will be tested for DTH to autologous NSCLC cells that have been: DNP-modified, or unmodified and irradiated, or unmodified and irradiated and fixed with ethanol (if sufficient cells available) Three doses of vaccine will be tested: 5 x 105, 2.5 x 106, or 5 x 106 DNP-modified autologous NSCLC cells. An initial dose of DNP-modified autologous NSCLC cells* without Bacillus of Calmette and Guérin (BCG) followed by cyclophosphamide (CY) then weekly doses of DNP-modified autologous NSCLC tumor cells mixed with BCG for 6 weeks, and completed with one dose of DNP-modified autologous NSCLC tumor cells mixed with BCG as a 6-month booster, if adequate number of cells available.

* count determined prior to aliquoting for cryopreservation

Endpoints: Treatment-emergent and related adverse events, serious adverse events, and Grade 3 and 4 laboratory abnormalities for safety assessments

Other Parameters: · DTH skin reactions for assessing the induction of immune responses to DNP-modified and unmodified autologous NSCLC tumor cells· Survival· Exploratory analysis of in vitro studies of peripheral blood lymphocytes obtained from study subjects

Duration of Treatment: Up to 9 months

Duration of Subject Participation in Study: Three months from the patient's last vaccine

Duration of Follow-up: Survival information and disease status will be collected via phone or visit on a quarterly basis for each patient beginning 30 days after the last scheduled visit until the last patient has been followed for three months from his/her last vaccine

Number of Subjects Required to Meet Protocol Objectives: Up to 42 evaluable subjects

Number of Study Centers: Three

Number of Individual Blood Draws: 15 draws over nine months

Volume of Blood Drawn: 13 Draws of 30 mL/draw (total 360 mL) and two draws of 50mL in heparinized tubes

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented stage IA, IB, IIA, IIB or IIIA NSCLC that is completely resectable and does not require post-operative radiation therapy or peri-operative chemotherapy
* Excision of the tumor and harvesting of tumor mass yielding adequate cells for vaccine manufacture and DTH testing
* Successful preparation and lot release of vaccines and of DTH testing material containing DNP-modified tumor cells
* Minimum of 3 and maximum of 8 weeks since the surgery
* Expected survival of at least 6 months
* Karnofsky performance status ³ 80
* Signed informed consent

Exclusion Criteria:

Alkaline phosphatase > 2.5 x ULN

* Total bilirubin > 2.0 mg/dL
* Creatinine > 2.0 mg/dL
* Hemoglobin < 10.0 g/dL
* WBC < 3,000 /mm3
* Platelet count < 100,000/mm3
* Chemotherapy - pre-operative or post-operative (except as designated in protocol)
* Radiation therapy to lung - pre-operative or post-operative
* Any major field radiotherapy within 6 months prior to participation in the study
* Immunotherapy (interferons, tumor necrosis factor, other cytokines [e.g., interleukins], biological response modifiers, or monoclonal antibodies) within 4 weeks prior to participation in the study
* Prior splenectomy
* Concurrent use of systemic steroids, except for the period of administration of the adjuvant chemotherapy, as per Section 8.6 (months 4-7)(Note: Topical steroid therapies [applied to the skin] are allowed, provided these are not applied to limbs injected with vaccine or skin test materials. Inhaled aerosol steroids are allowed.)
* Concurrent use of immunosuppressive drugs, except for the period of administration of the adjuvant chemotherapy (months 4-7)
* Concurrent use of antitubercular drugs (isoniazid, rifampin, streptomycin)
* Other malignancy within 5 years except curatively treated non-melanomatous skin cancer and curatively treated carcinoma in situ of the uterine cervix, or early stage (stage A or B1) prostate cancer
* Concurrent autoimmune diseases, e.g., systemic lupus erythematosus, multiple sclerosis or ankylosing spondylitis
* Concurrent medical condition that would preclude compliance or immunologic response to study treatment
* Concurrent serious infection or other serious medical condition
* Receipt of any investigational medication within 4 weeks prior to participation in the study
* Pregnancy or lactation (serum b-human chorionic gonadotropin [b-HCG] test must be negative in fertile women at screening visit)
* Active tuberculosis or a past history of tuberculosis
* PPD positive (³ 5 mm to 5TU)
* Known gentamicin sensitivity
* Anergic, defined by the inability to make a DTH to at least one of the following: candida, mumps, tetanus or trichophyton (based, except for the period of administration of the adjuvant chemotherapy (months 4-7) upon availability)
* Vaccine lot release failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cell-mediated immunity to autologous tumor cells. | 3 months
Safety | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Henry E Schea, Study Director — AVAX Technologies
Locations (2):
- United States (2):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Berd D, Sato T, Cohn H, Maguire HC Jr, Mastrangelo MJ. Treatment of metastatic melanoma with autologous, hapten-modified melanoma vaccine: regression of pulmonary metastases. Int J Cancer. 2001 Nov;94(4):531-9. doi: 10.1002/ijc.1506.abs. PMID 11745440